CLINICAL TRIAL: NCT01638299
Title: Feasibility Study Assessing the Ability of an Insulin Pump-controlling Algorithm to Minimize Hypoglycemia and Hyperglycemia in Patients With Type 1 Diabetes in a Clinical Research Setting
Brief Title: Study Assessing an Insulin Pump-controlling Algorithm to Minimize Hypo and Hyper in Type 1 During CRC Setting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Animas Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3076823, V3.0
Record Dates: First submitted 2012-06-25; First posted 2012-07-11 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; Artificial Pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypo-Hyper Minimizer (HHM) System (Experimental)
  Interventions: Device: Hypo-Hyper Minimizer (HHM) System

INTERVENTIONS:
Device: Hypo-Hyper Minimizer (HHM) System — Adjustment of Insulin dosing during meal time
  Other Names: Insulin delivery

SUMMARY:
Feasibility study assessing the ability of an insulin pump-controlling algorithm to minimize hypoglycemia and hyperglycemia in patients with type 1 diabetes in a clinical research setting.

DETAILED DESCRIPTION:
This study is a non-randomized, uncontrolled feasibility study that looks to enroll people with type 1 diabetes who are currently using an insulin pump. During the subject's participation, the study staff will closely monitor the study subject in a clinical research center environment for approximately 30 hours, while controller algorithm determined insulin doses are delivered by an insulin pump, and utilizing continuous glucose monitoring results.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-65 years
* type 1 diabetes mellitus for at least one year
* Currently using an insulin infusion pump for at least the past 6 months

Exclusion Criteria:

* Pregnancy
* History of Diabetic Ketoacidosis (DKA) in the past six months
* Histoey of severe hypoglycemia (Seizure, unconsciousnesss) in the past 6 months

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the performance of the HHM system response to meal insulin while the subject is under close medical supervision in the Clinical Research Center (CRC) setting. | After subject is discharged from CRC, 1 week after enrolment

SECONDARY OUTCOMES:
Number of Safety Events and any additional information that can be used for product development | After subject is discharged from CRC, 1 week after enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Henry Anhalt, DO, Study Director — Animas Corporation
Locations (2):
- United States (2):
  - Samsum Diabetes Reserach Inst., Santa Barbara, California
  - UVA Diabetes Technology Center, Charlottesville, Virginia